CLINICAL TRIAL: NCT02466230
Title: Predictive and Response Biomarkers of Effective Treatment With Transcranial Magnetic Stimulation for Major Depressive Disorder
Brief Title: Antidepressant Mechanisms of Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1101011475
Record Dates: First submitted 2015-05-28; First posted 2015-06-09 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Depression
Keywords: Magnetic stimulation of the brain; Antidepressant mechanisms
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active rTMS (Experimental): Subjects in the active rTMS arm will receive daily active repetitive transcranial magnetic stimulation (rTMS) treatments for 25 days (Monday through Friday for 5 consecutive weeks). Active rTMS with the FDA approved Neuronetics TMS system will be administered. Each treatment will target the left dorsolateral prefrontal cortex. rTMS will be administered at 10Hz with a duty cycle of 4 seconds on and 26 seconds off for 37.5 min.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Active repetitive transcranial magnetic stimulation for 25 days (Monday through Friday for 5 consecutive weeks). Active rTMS with the FDA approved Neuronetics TMS system. Each treatment will target the left dorsolateral prefrontal cortex. rTMS will be administered at 10Hz with a duty cycle of 4 seconds on and 26 seconds off for 37.5 min.

SUMMARY:
This study utilizes resting state fMRI, arterial spin labelling imaging, diffusion tensor imaging, structural MR-imaging, and MR-spectroscopy of GABA and Glutamate to probe the antidepressant mechanisms of repetitive transcranial magnetic stimulation (rTMS). The above imaging modalities will be acquired before and after an open-label 5 week course of rTMS for depression in currently depressed individuals with treatment resistant depression. Changes in functional, structural, and neurochemical markers will be investigated in rTMS responders and nonresponders to elucidate mechanisms of plasticity that correlate with treatment response. Additionally, functional, structural, and neurochemical signatures at baseline that correlate with subsequent treatment response will be investigated.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) applied over the left dorsolateral prefrontal cortex (DLPFC) alleviates mood in major depression. This treatment received FDA approval in 2009 and is now in routine clinical use for the treatment of major depression. A recently published sham-controlled study showed a response rate of 14% in real rTMS compared to 5% in sham rTMS. The response, defined by a greater than 50% reduction in the Hamilton Depression Rating Scale from pre-treatment to post-treatment, was also found to be 14% in one recent meta-analysis. The inclusion criteria in these studies admitted a broad spectrum of participants, ranging from subjects having a first major depressive episode, to those having failed multiple medication trials, suggesting that a subgroup with a more robust response may be masked by an unresponsive group. Abnormal function of the left frontal lobe accompanies major depression and this may be normalized by rTMS Cerebral blood flow measured with SPECT imaging was reduced in the left DLPFC of depressed subjects and was increased during and after a course of rTMS over the left DLPFC. Decreased blood flow was found in a broader region of frontal and paralimbic regions in depressed individuals and treatment success was associated with decreased blood flow in the inferior frontal lobes both pre- and post- treatment. Greater post-treatment vs. pre-treatment BOLD activation of left frontal regions was demonstrated using fMRI in a planning task that engages the frontal lobes. Left prefrontal myo-inositol is reduced in depressed subjects and this is normalized by rTMS. The above functional abnormalities view the frontal lobe in isolation. However, recent work has demonstrated a network-based structural marker of risk for familial depression consisting of decreased cortical and white mater volume. Resting state fMRI (rs-fMRI) tests cross-regional temporal coherence in low frequency oscillations in brain responses (~0.1 Hz) that are believed to represent spontaneous neural activity. Correlated spontaneous fluctuations are understood to reflect functional connections between brain regions that arise through a history of co-activation across one's lifetime. Previous work has shown that depressed patients exhibit altered functional connectivity patterns as gauged by rs-fMRI, and some studies suggest that these differences may be mitigated by treatment with antidepressant medications. However, whether and how TMS may affect functional connectivity is unknown. I propose to acquire the several described MRI types both before and after rTMS treatment in a search for predictive markers of rTMS treatment success as well as markers of treatment-induced change. Arterial spin labeling will be acquired to measure the blood flow distribution throughout the brain, both to confirm the SPECT results already reported and to test for additional regions of change. Resting state fMRI will be collected and DTI will be used to explore the structural basis of functional network changes. Structural MRI will be collected to measure cortical thickness and white matter volumes that may be predictive of rTMS response. Magnetic resonance spectroscopy will be collected to confirm the previously reported finding of rTMS-induced myo-inositol changes, as well as to consider the Glutamate/Glutamine and GABA spectra, given the importance of these neurotransmitters in theories of depression.

ELIGIBILITY:
Inclusion Criteria:

1. A history of major depressive disorder by the Structured Clinical Interview for DSM-IV (SCID)
2. Failure to respond to at least two previous antidepressant trials at adequate doses for 8 weeks (for current or prior major depressive episodes)
3. A minimum 17-item Hamilton depression rating scale of 17 on both the screening day and the treatment day #1
4. Age 18-70
5. Participants may be taking antidepressants, antipsychotics, or low-dose mood stabilizers during the study
6. Participants may be in psychotherapy during the study

Exclusion Criteria:

1. Participants with metal implants (Will use the NY Presbyterian Hospital MRI Checklist)
2. Prior exposure to TMS
3. Pregnant women
4. Lactating women
5. Bipolar disorder (on the Structured Clinical Interview for DSM-IV (SCID)
6. Current depressive episode longer than 3 years
7. Active suicidal ideation with plan or intent
8. Borderline personality disorder (on the Structured Clinical Interview for DSM-IV (SCID)
9. Substance abuse or dependence with the past 3 years
10. Current urine drug screen positive for any drugs of abuse
11. Current symptoms of psychosis
12. History of seizure disorder
13. History of closed head injury with loss of consciousness
14. History of brain surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Dubin, MD, PhD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant Flow of the Overall Study.
Pre-assignment Details: 28 subjects were enrolled and all completed the study.
Period: Overall Study
Arm/Group | Active rTMS
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active rTMS
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
Hamilton Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale is 24 items with total scores ranging from 0-76. Higher scores indicate greater severity of depression. (0-7 = None; 8-13 = Mild; 14-18 = Moderate; 19-23 = Severe; 23 and higher = very severe). Total scores are reported with no subscales.
  units on a scale | 27.6 (6.5)
Patient Health Questionnaire - 9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Self-rated scale of symptoms of depression. Nine items with a maximum score of 27. Higher score means more severe depression (0-4 = None; 5-9 = Mild; 10-14 = Moderate; 15-19 = Severe; 20 and higher = Very Severe).
  units on a scale | 14.3 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity Measured by the Hamilton Depression Rating Scale (24-Item)
Description: The Hamilton Depression Rating Scale is 24 items with total scores ranging from 0-76. Higher scores indicate greater severity of depression. (0-7 = None; 8-13 = Mild; 14-18 = Moderate; 19-23 = Severe; 23 and higher = very severe). Total scores are reported with no subscales.
Time Frame: Change in score on Hamilton Depression Rating Scale from baseline to immediately after the final rTMS treatment (5 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS
Number analyzed (Participants) | 28
units on a scale | 18.2 (7.7)

2. Secondary Outcome: Depression Severity Measured by the Public Health Questionnaire-9
Description: Self-rated scale of symptoms of depression. Nine items with a maximum score of 27. Higher score means more severe depression (0-4 = None; 5-9 = Mild; 10-14 = Moderate; 15-19 = Severe; 20 and higher = Very Severe).
Time Frame: Change in score in Public Health Questionnaire-9 from baseline to immediately after the final rTMS treatment (5 weeks)
Population: All 28 subjects completed the study but two subjects did not complete the final PHQ-9 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS
Number analyzed (Participants) | 26
units on a scale | 9.7 (6.3)

3. Other Pre Specified Outcome: Gamma-amino-butyric Acid Level Measured by Magnetic Resonance Spectroscopy
Description: Percent change in medial prefrontal gamma-amino-butyric acid level
Time Frame: Baseline to immediately after the final rTMS treatment (5 weeks)
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Glutamate Level Measured by Magnetic Resonance Spectroscopy
Description: Percent change in medial prefrontal glutamate level
Time Frame: Baseline to immediately after the final rTMS treatment (5 weeks)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Cortical Thickness Measured by T1 Magnetic Resonance Imaging
Description: Percent change in medial prefrontal average cortical thickness
Time Frame: Baseline to immediately after the final rTMS treatment (5 weeks)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Fractional Anisotropy Measured by Diffusion Tensor Imaging
Description: Percent change in medial prefrontal average fractional anisotropy
Time Frame: Baseline to immediately after the final rTMS treatment (5 weeks)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Functional Connectivity Measured by Functional Magnetic Resonance Imaging
Description: Percent change in medial prefrontal average functional connectivity
Time Frame: Baseline to immediately after the final rTMS treatment (5 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Five weeks (25 days)
Arm/Group | Active rTMS
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes